CLINICAL TRIAL: NCT02576171
Title: Group Therapy Supported Internet-based Cognitive Behavioral Therapy for Adolescents With Social Anxiety Disorder - A Feasibility Trial
Brief Title: Group Therapy Supported Internet-based CBT for Adolescents With Social Anxiety Disorder - A Feasibility Trial
Acronym: SoFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Serlachius, Associate professor, child psychiatrist, MD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SoFT Pilot
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Social Anxiety Disorder
Keywords: cognitive behavioral therapy;; guided self-help; adolescent
MeSH Terms: conditions — Phobia, Social | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group-therapy + ICBT (Experimental): This is an open trial with only one study arm
  Interventions: Behavioral: Group-therapy + ICBT

INTERVENTIONS:
Behavioral: Group-therapy + ICBT — The group therapy supported ICBT treatment program is a combined web-based and face-to-face intervention that will involve adolescents as well as their parents. The program is founded on and inspired by previously evaluated and evidence-based interventions. Altogether, adolescents go through 12 chapters/sessions, 3 of which are face-to-face group sessions at the research clinic, and 9 of which are web-bases chapters. The program is divided into three different phases, starting with psychoeducation regarding social anxiety and the rationale for a cognitive behavioral intervention. Phase two is the main part of treatment and contains behavioral interventions, mainly exposure and habituation to feared situations and/or stimuli.

SUMMARY:
The primary objectives of this study is to test the feasibility and efficacy of group-therapy supported internet-delivered CBT for adolescents (13 - 17 years) with social anxiety disorder. Investigators will conduct an open trial with N = 30 participants. Participants will be assessed at baseline, immediately after treatment and at a 6-month follow-up.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) among youths is highly prevalent and causes significant impairment in the lives of the affected. In spite of CBT being the most effective treatment, evidence suggests that many young people with this disorder do not have access to good-quality CBT. Internet-based CBT is, as numerous prior studies have shown, an effective method to treat psychiatric conditions in adults, but little is known about ICBT for adolescents and there are but a few controlled studies on ICBT for children and adolescents with anxiety disorders. This pilot trial will evaluate the feasibility and efficacy of a blended ICBT-treatment where internet-based and group-based sessions are combined. Furthermore, as ICBT is a novel format in the treatment of psychological problems in young people, it is essential to evaluate the feasibility and acceptability of the technical solutions that carry the active treatment. The study will also include genotyping of participants to further our understanding of etiology of SAD and to explore the relationship between genetic variations and treatment outcome. Additionally, as there is little known about the affect of ASD symptoms on treatment outcome in face-to-face CBT in general, and in ICBT in particular, the association between autistic traits and treatment outcome will be evaluated. Lastly, the role of attentional processes in the maintenance of social anxiety has been scarcely studied and an aim with the current study is to further our understanding of the cognitive factors that underlie SAD

ELIGIBILITY:
Inclusion Criteria:

* A principal diagnosis of social anxiety disorder, as defined by DSM-5
* Ability to read and write Swedish
* Daily access to the internet through a computer or similar device
* A parent or caregiver that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* Diagnosed with autism spectrum disorder, psychosis, bipolar disorder or severe eating disorder
* Present risk of suicide
* Ongoing substance dependence
* Occurrence of domestic violence
* Completed CBT for any anxiety disorder within the last 6 months (defined as at least 5 sessions of CBT including in vivo exposure sessions)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression - Severity | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
  Change from Baseline of social anxiety disorder severity, after 12 weeks and at 6 months after treatment

SECONDARY OUTCOMES:
Presence of DSM-5 Social Anxiety Disorder | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
Clinical Global Impression - Improvement | Assessed 12 weeks after treatment starts and 6 months after treatment has ended
Social Phobia and Anxiety Inventory (SPAI) - Child version | Assessed at baseline, Mid-3 weeks, Mid-6 weeks, Mid-9 weeks, 12 weeks after treatment starts and 6 months after treatment has ended
Social Phobia and Anxiety Inventory (SPAI) - Parent version | Assessed at baseline, Mid-3 weeks, Mid-6 weeks, Mid-9 weeks, 12 weeks after treatment starts and 6 months after treatment has ended
Revised Children´s Anxiety and Depression Scale (RCADS) - Child version | Assessed at baseline, Mid-6 weeks, 12 weeks after treatment starts and 6 months after treatment has ended
Revised Children´s Anxiety and Depression Scale (RCADS) - Parent version | Assessed at baseline, mid-6 weeks, 12 weeks after treatment starts and 6 months after treatment has ended
Children's Global Assessment Scale (CGAS) | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
Social Phobia Weekly Summary Scale (SPWSS) | Assessed at baseline, Mid-3 weeks, Mid-6 weeks, Mid-9 weeks, 12 weeks after treatment starts and 6 months after treatment has ended
Patient ICBT Adherence Scale (PIAS) | Assessed at Mid-6 weeks and 12 weeks after treatment starts
KIDSCREEN-10 - Child version | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
KIDSCREEN-10 - Parent version | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
Education, Work and Social Adjustment Scale - child version | Assessed at baseline, Mid-6 week, 12 weeks after treatment starts and 6 months after treatment has ended
Education, Work and Social Adjustment Scale - parent version | Assessed at baseline, Mid-6 week, 12 weeks after treatment starts and 6 months after treatment has ended
Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness - Child version (TiC-P) | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
Client Satisfaction Scale (CSS) | Assessed at 12 weeks after treatment starts
Measurement of anxiety levels during exposure (app) | Assessed from Mid-4 week to 12 weeks after treatment starts
Unintended treatment effects | Assessed at 12 weeks after treatment starts
  Open ended question where participants report any possible negative consequence of the treatment
Technology acceptance scale (TAS) - child version | Assessed at Mid-3 week and 12 weeks after treatment starts
Technology acceptance scale (TAS) - parent version | Assessed at Mid-3 week and 12 weeks after treatment starts
Hospital Anxiety and Depression Scale (HADS) | Assessed at baseline.
Social Responsiveness Scale - Parent version | Assessed at baseline.
DNA through saliva sampling | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
Attention bias when presented with social stimuli (eye-tracking) | Assessed at baseline, 12 weeks after treatment starts and 6 months after treatment has ended
Qualitative interviews of experience from treatment | Assessed at 12 weeks after treatment starts

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, Ass. Prof., Principal Investigator — Karolinska Institutet
Locations (1):
- BUP CPF, Stockholm, Sweden

REFERENCES:
- [Derived] Nordh M, Vigerland S, Ost LG, Ljotsson B, Mataix-Cols D, Serlachius E, Hogstrom J. Therapist-guided internet-delivered cognitive-behavioural therapy supplemented with group exposure sessions for adolescents with social anxiety disorder: a feasibility trial. BMJ Open. 2017 Dec 14;7(12):e018345. doi: 10.1136/bmjopen-2017-018345. PMID 29247101